CLINICAL TRIAL: NCT05396027
Title: Study of Effectiveness of Audio Guided Deep Breathing on Improving the Quality of Life of Physically Disabled Group
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Poh Foong Lee, PhD, Assistant Professor, Universiti Tunku Abdul Rahman
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IPSR/RMC/UTARRF/2020-C2/L05; IPSR/RMC/UTARRF/2020-C2/L05 (Other Grant/Funding Number: University Tunku Abdul Rahman)
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Psychophysiology; Visually Impaired Persons; Physiological Phenomena; Psychological Stress
Keywords: Guided Deep Breathing; Visual Impairment; Physical Disability; Mental Stress
MeSH Terms: conditions — Stress, Psychological; Vision Disorders

STUDY DESIGN:
Intervention Model Description: The crossover study design is implemented whereby healthy participants are assigned to the control group whereas visually impaired participants are assigned to the intervention group initially. After 14 days, the same participants cross over from the first session to the second session during the experiment.
Who Masked: Participant
Masking Description: Participants do not know which study group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants (healthy or physically disabled) in the control group do not require to perform audio-guided deep breathing for 14 days continuously
- Experimental Group with Audio-guided deep breathing (Experimental): Participants (healthy or physically disabled) in the interventional group need to perform 5 mins audio-guided deep breathing with 6 deep breaths per minute for 14 days continuously
  Interventions: Other: Audio-guided deep breathing

INTERVENTIONS:
Other: Audio-guided deep breathing — 2 weeks of audio-guided deep breathing for participants (healthy and physically disabled)
  Arms: Experimental Group with Audio-guided deep breathing

SUMMARY:
Diaphragmatic breathing brings different advantages to improve physical and mental health but it could be difficult for the physically disabled group to follow the practice by themselves especially those with vision impairment. Therefore, guided deep breathing is desirable to address their needs but these are rarely analyzed in the previous literature. This research aims to study the physiological impacts and psychological health of audio-guided deep breathing on physically disabled groups. The psychological changes will be assessed by Perceived Stress Scale (PSS), World Health Organization Quality of Life (WHO-BREF) and Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Besides, physiological parameters such as tidal volume, electroencephalography, hair cortisol level and heart rate variability are measured non-invasively to evaluate the impact of audio-guided deep breathing. Furthermore, auditory Go-No Go Task will be adopted as a neuropsychological test in determining changes in response control and sustained attention in this study as well. Eventually, the pre-and post-interventional data will be analyzed and processed to study the effect of audio-guided deep breathing on these special groups.

DETAILED DESCRIPTION:
Background:

Diaphragmatic breathing is also known as deep breathing as the breathing process is always associated with belly expansion, diaphragm contraction, and deep inhalation and exhalation which results in greater intake of blood gases and reduced respiratory frequency that is in contrast to the normal breathing cycle. Some of the studies revealed the potentiality of deep breathing in enhancing social adaption, emotional balance, stress management and physiological stability. The advantages of deep breathing also have been reported extensively in ancient eastern religions, including yoga, meditation and Tai Chi Chuan (TCC). The positive outcomes of deep breathing have evoked scientific interest in the investigation of the causal relationship between deep breathing practice and physiological behaviours. Since deep breathing is voluntary respiration which is opposed to natural breathing, it will give rise to certain degrees of physiological changes unavoidably. Physiological changes including tidal volume, heart rate variability, electroencephalography and hair cortisol level have been reported in the previous works of literature.

Literature Review:

Effect of Deep Breathing on Pulmonary Function

To achieve optimal oxygen saturation level, tidal volume and respiratory rate are the two primary components of respiratory measurement responsible for the purpose. Tidal volume is the amount of air-filled in each breathing cycle. Under relaxed conditions, these two parameters change interchangeably to optimize oxygen intake. Since deep breathing is involuntary breathing, it inevitably brings changes to the pulmonary parameters. For example, some researchers found out that tidal volume and other pulmonary parameters such as forced expiratory volume and forced vital capacity increased after ten minutes of deep breathing compared to normal chest breathing. Some authors also agreed that the deep breathing technique showed improvement in pulmonary function in a healthy subject.

Effect of Deep Breathing on Heart Rate Variability

Heart Rate Variability (HRV) is modulated by autonomic nervous system and further divided into two branches: sympathetic and parasympathetic pathways. The sympathetic nervous system is concerned with critical events such as respiratory failure and survival challenges that causes blood pressure and heart rate to increase. This is known as the "fight-or-flight" reaction. In contrast, the parasympathetic nervous system focuses on the resting and conservation of energy that acts in opposition to the sympathetic pathway. They work together dynamically giving rise to HRV and serving as a measurable index of autonomic control. It was reported that breathing can influence cardiopulmonary function that indirectly reflects HRV. Inhalation and exhalation alter the heart rate which is known as respiratory sinus arrhythmia (RSA). In other words, inhalation reduces R-R intervals in electrocardiogram (ECG) and increases during exhalation. Slow and deep breathing which has lower respiratory frequency is found to augment cardiorespiratory synchronization and elevate HRV. Most of the studies reported that slow and deep breathing can bring positive effects to HRV that is associated with stress, diabetes mellitus and rheumatoid arthritis.

The analysis of HRV can be divided into time-domain and frequency-domain analyses. In frequency-domain analysis, there are high-frequency spectrum (HF) (0.14 Hz - 0.40 Hz) and low-frequency spectrum (LF) (0.04 Hz - 0.15 Hz) that refer to parasympathetic and sympathetic activities respectively. On the other hand, time-domain analysis, for instance, root mean square of the variation in R-R interval (RMSSD), N-N interval standard deviation (SDNN) and average R-R intervals standard deviation (SDANN) are begin measured as the units.

One of the studies suggested that LF increased at once after five minutes of deep breathing whereas SDNN and RMSSD changes are insignificant. Conversely, a pilot study on the impact of different deep breathing duration reported showed that normalized HF power is smaller than the control group without deep breathing. This study suggested that depression score is lower in the deep breathing groups with lower HF reading. The difference is due to the sympathetic activation being involved when a novel and short exercise was provided whereas long training will shift to parasympathetic activation. Another research also suggested that SDNN increased after deep breathing indicating stress relief.

Effect of Deep Breathing on Electroencephalography (EEG)

Electroencephalography (EEG) is a well-known screening technique to acquire the scalp electrical behaviour of the brain. The electrical activity is a product of neuron activation in the brain that causes a flow of current. During the event of synaptic activation in the cerebral cortex, the current flow is the one captured by EEG. There have been numerous studies to investigate the application of EEG in neurology and neuropsychology studies due to its strong ability in receiving neurofeedback from the brain from the past until now.

The brainwave is classified into four mainly by the amplitude and frequency differences. Alpha waves (8 - 13 Hz) is associated with the mental task, awake or resting that is recorded in the parieto-occipital area. Next, beta waves (14 - 30 Hz) is gathered during mental activity similarly which is presented in the parietal or frontal region while theta waves (4 - 7 Hz) is found when an adult is sleeping or drowsy but it also indicates stress when the adult is waked. The last wave is delta waves (< 3.5 Hz) which shows that an adult is in deep sleep or severe brain damage in waked adult.

These brainwaves are shown to correlate with deep breathing. Alpha wave is associated with relaxation and stability while beta wave shows certain degrees of stress and stimulation. For example, it was suggested that slow and deep breathing elevated alpha to the high beta ratio which indicates improvement of mental stability. Similarly, deep breathing, as an important element in mediation and yoga practice also has proposed that it increased alpha power in prior studies. On the other hand, some studies showed that beta activity decreased after slow and deep breathing but some studies oppose the findings. Previous research projects have documented that frontal theta power increased is associated with reduced anxiety as well.

Effect of Deep Breathing on Cortisol Level

In the event of the stress response, a cascade reaction of hormone occurs at the pituitary gland, hypothalamus and adrenal gland. Glucocorticoids is a compound as a result of the stimulation play an important role in stress coping that could activate a series of physiological responses such as immune activation, inflammatory suppression, reproductive physiology reduction and energy mobilization. Hair cortisol analysis is a relatively novel technique compared to saliva and urine cortisol analysis. Although the mechanism of cortisol deposition is pending further investigation, it is a promising technique with more benefits. It is non-invasive, unlikely to be affected by sampling procedures, lower storage requirement and cortisol production measured has a longer timeframe (months to years). Therefore, it is considered a good biomarker of chronic stress level that has driven several studies such as antenatal stress, relaxation interventions, early childhood and neonates.

Deep breathing has been shown to reduce cortisol levels which were reported by previous studies. However, they were using saliva and plasma for the assessment respectively. Similarly, some authors have provided evidence of interventions that are incorporated with deep breathing reported to reduce cortisol levels as well. For example, it was suggested that laughter yoga that involved deep breathing as one of the components has shown a reduction in salivary cortisol levels. For hair cortisol assessment, one study used this technique that stress reduction program with deep breathing component proved that cortisol level was reduced. The relationship between hair cortisol and deep breathing intervention is rarely analyzed in the previous studies. A closer look at the literature on intervention incorporated with a deep breathing exercise, however, reveals a question of whether deep breathing alone was contributing to the reduction of hair cortisol. Therefore, this was an important question to study the effect of deep breathing exercise itself on hair cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Visual Acuity in the better-seeing eye worse than 6/12, according to the criteria of the World Health Organization (for visually impaired only).
* hair length of at least 1 cm long
* have consistent internet and computer/laptop/mobile phone access

Exclusion Criteria:

* fail to meet the above-listed inclusion criteria
* those who are unable to take deep breathing for 5 minutes or more
* having taken or on drug prescription and medication
* those who with a medical condition for the past two weeks other than visual impairment
* other long-term diseases or medical condition impacting physical disability
* those who do smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline stress by Perceived Stress Scale (PSS) | Baseline, 14 days
  PSS is an international instrument that is designed to evaluate the individual's stress level. It requires participants to rate their feeling and thoughts in the past month in the different cases provided. The rating is described as a scale of 0 (never) to 4 (very often). If the summated score is high, it is always associated with a higher level of perceived stress.
Change from baseline quality of life by World Health Organization Quality of Life - BREF (WHO-BREF) | Baseline, 14 days
  WHO-BREF consists of 26 items that are divided into four domains namely physical health, psychological, social relationships and environment to measure participants' quality of life. The scores follow five-point Likert Scales where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely". Higher scores indicate higher quality of life.
Change from baseline mindfulness level by Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Baseline, 14 days
  CAMS-R is a ten-item scales designed to measure one's mindfulness approach to relate their feeling, emotion and thought. It is presented in four Likert scales from 1 (Rarely/Not at all) to 4 (Almost always) which require the participant to rate how applicable each item is to them.
Change from baseline Alpha waves by Non-invasive electroencephalogram (EEG) | Baseline, 7 days, 14 days
  The 32- channel electrodes were placed in compliance with the International 10-20 System nomenclature. The increase or decrease in Alpha wave EEG recordings of the participants are recorded in eyes closed for 1 min
Change from baseline Beta waves by Non-invasive electroencephalogram (EEG) | Baseline, 7 days, 14 days
  The 32- channel electrodes were placed in compliance with the International 10-20 System nomenclature. The increase or decrease in Beta wave EEG recordings of the participants are recorded in eyes closed for 1 min
Change from baseline Theta waves by Non-invasive electroencephalogram (EEG) | Baseline, 7 days, 14 days
  The 32- channel electrodes were placed in compliance with the International 10-20 System nomenclature. The increase or decrease in Theta wave EEG recordings of the participants are recorded in eyes closed for 1 min
Change from baseline hair cortisol level by hair cortisol analysis | Baseline, 14 days
  Hair samples will be collected from the participants. Scissors and hair clips will be used to collect hair samples closed to the scalp surface. Each hair sample will be stored in an envelope and labelled with a unique identification code according to the protocol provided by the laboratory appointed. Hair cortisol will be weighted, disinfected and pulverized into fine hair powder. Extraction methods will be applied to the samples by incubation and extraction solvent. The concentration will be measured using a commercially available ELISA kit
Change from baseline tidal volume by digital spirometer. | Baseline, 7 days, 14 days
  An electronic digital spirometer will be used to measure tidal volume. The participant will need to breathe out through a one-way valve disposable mouthpiece attached to the spirometer.
Change from baseline heart rate variability (HRV) by mobile HRV measurement software | Baseline, Day 1 to day 14
  A mobile HRV measurement software will be applied to measure the HRV of each participant. HRV Changes will be taken after the intervention for 14 days continuously.
  Change = (Day 14 - baseline, Day 7 - baseline, progressive changes (Day 1 - 14))
Change from baseline by Rosenberg's Self-Esteem Scale | Baseline, 14 days
  Rosenberg's Self-esteem scale is a ten-item scale designed to measure one's positive and negative values towards themselves. In other words, it is used to measure individual self-esteem. All answers are in 4-Likert Scales format from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicate higher self-esteem.

SECONDARY OUTCOMES:
Change in Go/no-go task performance assessed by the Auditory Go/no-go task | Baseline, 14 days
  Performance on go/no-go task as measured by reaction time, omission error, commission error and reaction time variability

CONTACTS AND LOCATIONS:
Locations (1):
- Tunku Abdul Rahman University, Cheras, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Based on informed consent, participants data not shared